CLINICAL TRIAL: NCT03518515
Title: Potato Consumption and Energy Balance: a Randomized, Controlled, Clinical Trial
Brief Title: Potato Consumption and Energy Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Alliance for Potato Research and Education (Other); Indiana University (Other)
Responsible Party: Principal Investigator, Daniel L. Smith, Jr., Co-Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB-300001187
Record Dates: First submitted 2018-04-24; First posted 2018-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Obesity
Keywords: nutrition intervention; potato consumption; energy balance
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- White potato (French fries) (Experimental): Participants will be asked to consume 1 serving of French fries each day for 30 days.
  Interventions: Other: White potato (french fries)
- White potato (French fries), +seasoning (Experimental): Participants will be asked to consume 1 serving of French fries with added seasoning each day for 30 days.
  Interventions: Other: White potato (French fries), +seasoning
- Almond (Active Comparator): Participants will be asked to consume 1 serving of almonds (calorie-matched to other arms) day for 30 days.
  Interventions: Other: Almond

INTERVENTIONS:
Other: White potato (french fries) — If randomized to this group, participants will be asked to consume 1 serving of French fries (~300 kcal) each day for 30 days as a part of their usual dietary intake. French fries will be portioned and provided to participants.
  Arms: White potato (French fries)
Other: White potato (French fries), +seasoning — If randomized to this group, participants will be asked to consume 1 serving of French fries (~300 kcal) with added potential glycemia modifying seasoning mix each day for 30 days as a part of their usual dietary intake. French fries and seasoning will be portioned and provided to participants.
  Arms: White potato (French fries), +seasoning
Other: Almond — If randomized to this group, participants will be asked to consume 1 serving of almonds that is calorically-matched to the French fries (~300 kcal) serving in the other arms each day for 30 days as a part of their usual dietary intake. Almonds will be portioned and provided to participants.
  Arms: Almond

SUMMARY:
A randomized, clinical trial will be performed to assess changes in body weight and fat mass with daily potato consumption versus a calorie-matched snack of almonds.

DETAILED DESCRIPTION:
This is a 30-day randomized, controlled trial with 3 arms: 1) non-potato food (almonds), 2) standard white potato French fry, 3) standard white potato French fry with potential glycemia-modulating spice/seasoning mix added.

Free-living study participants will be assigned to consume one of the 3 foods (calorie matched) each day for a 30-day period. Body composition (via dual energy x-ray absorptiometry; DXA), and blood chemistry will be assayed at baseline and study completion, along with a sub-sample of subjects participating in a meal-based tolerance tests at study completion.

ELIGIBILITY:
Inclusion Criteria:

* 18- 50 years old
* Body mass index (BMI) 20- 35
* No dietary restrictions or allergies
* Weight stable
* Access to camera through smartphone, computer or tablet

Exclusion Criteria:

* Pregnancy or anticipating pregnancy or lactation
* Nut or food allergy
* Diagnosed diabetes (Type 1 or 2)
* History of weight control surgery (bariatric or liposuction)
* Consumes >1 serving of potatoes daily before enrollment
* Weight loss or gain >5% within past 6 months
* Medical conditions or medications that would prevent the ability to comply with treatment assignment and/or affect energy balance
* Dependence on others for food procurement or preparation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
Change in fat mass | baseline and study completion (30 days)
  Determined by dual-energy X-ray absorptiometry.

SECONDARY OUTCOMES:
Change in body weight | baseline and study completion (30 day)
Change in fasting glucose | baseline and study completion (30 day)
Change in fasting insulin | baseline and study completion (30 day)
Change in HbA1c | baseline and study completion (30 day)
Change in caloric Intake | baseline and study completion (30 days)
  Dietary recall by 3 day food record.
Meal Tolerance Test | Study Completion (30 day)
  A subset of subjects from each diet group will participate in a meal-based tolerance test with the study food items.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Smith, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Smith DL, Hanson RL, Dickinson SL, Chen X, Goss AM, Cleek JB, Garvey WT, Allison DB. French-fried potato consumption and energy balance: a randomized controlled trial. Am J Clin Nutr. 2022 Jun 7;115(6):1626-1636. doi: 10.1093/ajcn/nqac045. PMID 35179193